CLINICAL TRIAL: NCT01102439
Title: Randomized, Factorial Study to Explore Interaction Between Aspirin and Clopidogrel in Stable Patients With Previous Myocardial Infarction or Coronary Artery Stent
Brief Title: Clopidogrel/Aspirin Interaction Study
Acronym: INTERACTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, John Eikelboom, MD., Population Health Research Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 10-082
Record Dates: First submitted 2010-04-08; First posted 2010-04-13 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease
Keywords: Clopidogrel; Aspirin; Interaction
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Standard dose clopidogrel (Active Comparator): 300 mg Loading x 1 day, 75 mg/d x 13 days
  Interventions: Drug: Clopidogrel
- Double dose clopidogrel (Experimental): 600 mg Loading x 1 day, 150 mg/d x 6 days, 75 mg/d x 7 days
  Interventions: Drug: Clopidogrel
- Standard dose aspirin (Active Comparator): Aspirin 81mg/d x 14 days
  Interventions: Drug: Aspirin
- High dose aspirin (Experimental): Aspirin 325 mg/d x 14 days
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Clopidogrel — 300 mg loading dose, then 75 mg daily
  Other Names: Plavix
  Arms: Standard dose clopidogrel
Drug: Clopidogrel — 600 mg loading dose, 150 mg daily day 2-7, then 75 mg daily
  Other Names: Plavix
  Arms: Double dose clopidogrel
Drug: Aspirin — 81 mg daily
  Other Names: Entrophen
  Arms: Standard dose aspirin
Drug: Aspirin — 325 mg daily
  Other Names: Novasen
  Arms: High dose aspirin

SUMMARY:
This study will explore the effect of different doses of aspirin on the effects of double-dose or standard dose clopidogrel.

DETAILED DESCRIPTION:
Study Hypothesis: Patients receiving double-dose compared with standard-dose clopidogrel will have increased blood concentrations of the active metabolite of clopidogrel and greater inhibition of ADP-induced platelet aggregation when also treated with acetylsalicylic acid (ASA) 325 mg/d as compared to ASA 81 mg/d.

ELIGIBILITY:
Inclusion Criteria:

* > 1 month post myocardial infarction (MI), unstable angina or stent patients with stable condition
* Receiving regular ASA (81mg/d) and clopidogrel (75mg/d) for at least 1 week
* Written informed consent

Exclusion Criteria:

* Age < 18 years old
* Liver disease with transaminases and/or bilirubin > 1.5x upper limits of normal (ULN) (within 3 months of randomization)
* Renal impairment with creatinine clearance < 30 ml/min (within 3 months of randomization)
* Platelet count < 100x109/L and/or Hb< 100g/L (within 3 months of randomization)
* Use of oral anticoagulants or nonsteroidal antiinflammatory drug (NSAID) within the last 10 days or planned use during the study
* Use of antiplatelet agent other than aspirin and clopidogrel within the last 10 days
* High risk of bleeding (e.g. recent gastrointestinal bleeding, bleeding diathesis)
* Uncontrolled hypertension (> 180/110mmHg)
* Current smoker with ≥ 5 cigarettes/day
* Previously entered in this study or just finished other study within 2 weeks before recruitment
* Medical, geographic, or social factors making study participation impractical, or inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Blood concentrations of the active metabolite of clopidogrel | 14 days

SECONDARY OUTCOMES:
Inhibition of adenosine diphosphate (ADP) induced platelet aggregation | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liang, MD, Principal Investigator — Population Health Research Institute; John Eikelboom, MD., Study Director — Population Health Research Institute
Locations (1):
- Population Health Research Institute, Hamilton, Ontario, Canada